CLINICAL TRIAL: NCT01504191
Title: A Randomized Controlled Study of the Effects of Internet-based Cognitive Behavior Therapy on Depression and Anxiety in Patients With a Previous Myocardial Infarction
Brief Title: Internet-based Cognitive Behavior Therapy After Myocardial Infarction
Acronym: U-CARE: Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Louise-von Essen, Programme Director for U-CARE, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U-CARE: Heart
Record Dates: First submitted 2011-12-19; First posted 2012-01-05 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Depression; Anxiety; Myocardial Infarction
Keywords: myocardial infarction; depression; anxiety; Internet-based CBT; genetic disposition
MeSH Terms: conditions — Depression; Anxiety Disorders; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based CBT (Experimental): Randomized patients with symptoms of anxiety and/or depression after MI will participate in an Internet-based CBT-program.
  Interventions: Behavioral: Internet-based CBT
- Treatment as usual (TAU) (No Intervention): Control: After randomization patients with symptoms of anxiety and/or depression after MI will participate in the treatment as usual (TAU).
  Reference: A reference group without depressive or anxiety symptoms will participate in the treatment as usual (TAU).

INTERVENTIONS:
Behavioral: Internet-based CBT — The participants read texts and do weekly homework assignments instructed from an Internet page. Additional resources like discussion forum, pictures, animations, videos and sounds will be a part of the treatment program.
  A psychologist will communicate with the participants through internal text-messages. The therapist will devote about 10 minutes to each participant each week via the Internet. The content of the intervention will be standard components from CBT, for example relaxation training, behavioral activation, exposure for fear related stimuli, cognitive restructuring, behavioral sleep treatment etc.
  Arms: Internet-based CBT

SUMMARY:
The overall aim and primary objective is to evaluate the effects on level of depression and anxiety of an Internet-based CBT-program in depressed and/or anxious patients after a myocardial infarction (MI).

DETAILED DESCRIPTION:
Major or minor depressive disorders and anxiety disorders are present in many patients with cardiovascular disease (CVD) and are associated with adverse cardiovascular outcomes, even after controlling for other risk factors. 500 patients with symptoms of anxiety and/or depression after MI will be randomized either to a 14 week Internet-based CBT-program or to treatment as usual (TAU) which is the control condition. A reference group of 250 participants without depressive or anxiety symptoms will also be studied during TAU. Data will be collected before, after and 7 months after treatment. Anxiety and depression according to ratings on the Hospital Anxiety and Depression Scale (HADS) are the primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients younger than 75 years with a recent acute MI (< 3 months)
* Depression and/or anxiety score of > 7 on one or both of the HADS subscales (concerns only the intervention, not the reference group)

Exclusion Criteria:

* Patients that are scheduled for a coronary artery bypass surgery (CABG)
* Unable or unwilling to use computer or Internet
* Difficulties in reading or understanding Swedish
* A life expectancy of less than a year
* Anticipated poor compliance (multi-disease, substance abuse etc.)
* Highly depressed or suicidal (MADRS-score > 29 or MADRS item 9 > 3)

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2013-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Depression (difference between the intervention and the control group) | At baseline and 3 months later (after intervention)
  Hospital Anxiety and Depression Scale (HADS) - depression ratings;
  Montgomery Åsberg Depression Rating Scale (MADRS)
Change in Anxiety (difference between the intervention and the control group) | At baseline and 3 months later (after intervention)
  Hospital Anxiety and Depression Scale (HADS) - anxiety ratings

SECONDARY OUTCOMES:
Change in Quality of Life (difference between the intervention and the control group) | At baseline, during, after (3 months after baseline) and 7 months after treatment
  Ratings on EQ5d and Ladder of Life (LL)
Change in Perceived Social Support (difference between the intervention and the control group) | At baseline, after (3 months after baseline) and 7 months after treatment
  ENRICHED Social Support Inventory (ESSI)-ratings
Change in Stress behaviors (difference between the intervention and the control group) | At baseline, after (3 months after baseline) and 7 months after treatment
  Everyday Life Stress Scale (ELSS)-ratings
Change in Fatigue (difference between the intervention and the control group) | At baseline, after (3 months after baseline) and 7 months after treatment
  Maastricht Questionnaire (MQ)-ratings
Change in Cardiac Anxiety (difference between the intervention and the control group) | At baseline, after (3 months after baseline) and 7 months after treatment
  Cardiac Anxiety Questionnaire (CAQ)-ratings
Change in Sleeping Problems (difference between the intervention and the control group) | At baseline, after (3 months after baseline) and 7 months after treatment
  Insomnia Severity Index (ISI)-ratings
Change in Posttraumatic Stress (difference between the intervention and the control group) | At baseline, after (3 months after baseline) and 7 months after treatment
  Posttraumatic Stress Disorder Checklist- Civilian Version (PCL-C)-ratings
Change in Posttraumatic Growth (difference between the intervention and the control group) | At baseline, after (3 months after baseline) and 7 months after treatment
  The Posttraumatic Growth Inventory - Short Form (PTGI-SF)-ratings
Quality of the Intervention | At baseline, after (3 months after baseline) and 7 months after treatment
  Behavioral Activation for Depression Scale (BADS)-ratings
Change to Follow-up in Anxiety (difference between the intervention and the control group) | At baseline, after (3 months after baseline) and 7 months after treatment
  Hospital Anxiety and Depression Scale (HADS) - anxiety ratings
Change to Follow-up in Depression (difference between the intervention and the control group) | At baseline, after (3 months after baseline) and 7 months after treatment
  Hospital Anxiety and Depression Scale (HADS) - depression ratings;
  Montgomery Åsberg Depression Rating Scale (MADRS)

CONTACTS AND LOCATIONS:
Overall Officials: Louise von Essen, PhD, Principal Investigator — Uppsala University
Locations (25):
- Sweden (25):
  - Ängelholms sjukhus, Ängelholm
  - Enköpings lassarett, Enköping
  - Falu Lasarett, Falun
  - Gävle sjukhus, Gävle
  - Sahlgrenska sjukhuset, Gothenburg
  - Hässleholms sjukhus, Hässleholm
  - Blekinge sjukhus, Karlskrona
  - Karlstad sjukhus, Karlstad
  - Kungälvs sjukhus, Kungälv
  - Skaraborgs sjukhus, Lidköping
  - Ljungby lasarett, Ljungby
  - Skånes universitetssjukhus, Malmo
  - Mora lassarett, Mora
  - Nyköpings sjukhus, Nyköping
  - Oskarshamns sjukhus, Oskarshamn
  - Universitetssjukhuset Örebro, Örebro
  - Piteå älvdals sjukhus, Piteå
  - Danderyds sjukhus, Stockholm
  - Karolinska sjukhuset i Huddinge, Stockholm
  - Karolinska sjukhuset i Solna, Stockholm
  - Södersjukhuset, Stockholm
  - Länssjukhuset Sundsvall-Härnösand, Sundsvall
  - Uppsala Akademiska sjukhus, Uppsala
  - Varberg sjukhus, Varberg
  - Växjö centrallasarett, Vaxjo

REFERENCES:
- [Derived] Leissner P, Held C, Rondung E, Olsson EMG. The factor structure of the cardiac anxiety questionnaire, and validation in a post-MI population. BMC Med Res Methodol. 2022 Dec 29;22(1):338. doi: 10.1186/s12874-022-01820-5. PMID 36581833
- [Derived] Humphries SM, Wallert J, Norlund F, Wallin E, Burell G, von Essen L, Held C, Olsson EMG. Internet-Based Cognitive Behavioral Therapy for Patients Reporting Symptoms of Anxiety and Depression After Myocardial Infarction: U-CARE Heart Randomized Controlled Trial Twelve-Month Follow-up. J Med Internet Res. 2021 May 24;23(5):e25465. doi: 10.2196/25465. PMID 34028358
- [Derived] Wallert J, Gustafson E, Held C, Madison G, Norlund F, von Essen L, Olsson EMG. Predicting Adherence to Internet-Delivered Psychotherapy for Symptoms of Depression and Anxiety After Myocardial Infarction: Machine Learning Insights From the U-CARE Heart Randomized Controlled Trial. J Med Internet Res. 2018 Oct 10;20(10):e10754. doi: 10.2196/10754. PMID 30305255
- [Derived] Norlund F, Wallin E, Olsson EMG, Wallert J, Burell G, von Essen L, Held C. Internet-Based Cognitive Behavioral Therapy for Symptoms of Depression and Anxiety Among Patients With a Recent Myocardial Infarction: The U-CARE Heart Randomized Controlled Trial. J Med Internet Res. 2018 Mar 8;20(3):e88. doi: 10.2196/jmir.9710. PMID 29519777
- [Derived] Norlund F, Olsson EM, Burell G, Wallin E, Held C. Treatment of depression and anxiety with internet-based cognitive behavior therapy in patients with a recent myocardial infarction (U-CARE Heart): study protocol for a randomized controlled trial. Trials. 2015 Apr 11;16:154. doi: 10.1186/s13063-015-0689-y. PMID 25873137
- See also: U-CARE — http://www.u-care.uu.se/?languageId=1